CLINICAL TRIAL: NCT05542589
Title: Efficacy of Phenytoin Phonophoresis on Pressure Ulcer Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003632
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Pressure Ulcer
Keywords: Phenytoin; phonophoresis; pressure ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenytoin phonophoresis group (Experimental): The topical phenytoin will be applied on the head of ultrasound and is usually given for 5-10 minute sessions, three times per week and six weeks as a total treatment duration.
  Interventions: Other: Phenytoin phonophoresis
- sham phenytoin phonophoresis group (Sham Comparator): The topical phenytoin will be applied on the head of ultrasound (sham ultrasound) and is usually given for 5-10 minute sessions, three times per week and six weeks as total treatment duration.
  Interventions: Other: Sham phenytoin phonophoresis

INTERVENTIONS:
Other: Phenytoin phonophoresis — Phenytoin phonophoresis for 5-10 minute sessions, three times per week and six weeks as a total period treatment.
  Arms: Phenytoin phonophoresis group
Other: Sham phenytoin phonophoresis — Sham phenytoin phonophoresis for 5-10 minute sessions, three times per week and six weeks as a total period treatment.
  Arms: sham phenytoin phonophoresis group

SUMMARY:
Efficacy of phenytoin phonophoresis on pressure ulcer healing

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the therapeutic effect of phenytoin phonophoresis on the healing of pressure ulcers.

Subjects: Forty patients suffering from pressure ulcers will be randomly divided into two equal groups each one has 20 patients, they will be selected from Al Kaser Al Aini. In this study, the patients will be randomly assigned into two equal groups (20 patients for each group) and will receive the treatment program three sessions per week for 6 weeks as a total period of treatment.

Phenytoin phonophoresis group (Study group): This group includes 20 patients with pressure ulcers who will receive topical phenytoin with ultrasound in addition to their conventional treatment.

Phenytoin phonophoresis group (Control group): This group will include 20 patients with pressure ulcers who will receive phenytoin with a placebo ultrasound.

Equipment and tools:

Measurement equipment: Saline injection method. Therapeutic equipment: Ultrasonic device, topical phenytoin, and hydrogel sheet.

ELIGIBILITY:
Inclusion Criteria:

Ages range from 40 to 60 years, both genders, patients with pressure ulcers, and patients who will sign their informed consent.

Exclusion Criteria:

Patients with a history of hypersensitivity to phenytoin, pneumonia, immune deficiency, infection, advanced diabetic patients, radiotherapy in the ulcer area, osteomyelitis in the ulcer area, venous ulcers, burn wounds, leprosy trophic ulcers, traumatic wounds, pregnant subjects, terminally ill subjects, and the use of antineoplastic agents or systemic glucocorticosteroids.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Change in wound volume | Baseline and six weeks after the intervention
  by saline gel injection method
  Amount of saline gel will be applied by steralized single use syringe in wound cavity then score this amount Amount of saline gel will be applied by steralized single use syringe in wound cavity then score this amount
  Amount of saline gel will be applied by steralized single use syringe in wound cavity then score this amount .

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa MA Elsayeh, PhD, Study Director — Cairo University
Locations (1):
- Shaimaa Mohamed Ahmed Elsayeh, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No